CLINICAL TRIAL: NCT06077396
Title: Does Radial Artery Cannulation Affect the Perfusion Index of the Hand in Liver Transplant?
Brief Title: Does Radial Artery Cannulation Affect the Perfusion Index(PI) of the Hand in Liver Transplant Operations?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, DUYGU DEMİROZ, Principal Investigator, Inonu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LIVER TRANSP
Record Dates: First submitted 2023-08-25; First posted 2023-10-11 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Perfusion; Complications; Arterial Catheterization, Peripheral
Keywords: perfusion index; liver transplantation; radial artery cannulation

STUDY DESIGN:
Intervention Model Description: Patients who underwent radial artery cannulation in liver transplantation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- To evaluate the effect of radial artery cannulation on hand perfusion (Other): To evaluate the effect of radial artery cannulation on hand perfusion
  Interventions: Procedure: radial artery cannulation

INTERVENTIONS:
Procedure: radial artery cannulation — radial artery cannulation

SUMMARY:
radial artery cannulation is performed by an experienced person, non-invasive blood pressure measurement will be made at 3 stages of the operation (dissection, anhepatic, neohepatic) and the effects of radial artery cannulation on the perfusion index will be evaluated by recording the correlation between radial artery and invasive measurements and the perfusion indexes of both hands simultaneously with Masimo.

DETAILED DESCRIPTION:
Arterial lines placement is for real-time monitoring of blood pressures and arterial blood sampling in critically ill patients or those undergoing complex procedures and surgeries.

Routine monitoring will be performed after the patients are taken to the operating room. Before bilateral radial artery cannulation, allen test will be performed and entrance perfusion indexes will be checked. After radial artery cannulation is performed by an experienced person, non-invasive blood pressure measurement will be made at 3 stages of the operation (dissection, anhepatic, neohepatic) and the effects of radial artery cannulation on the perfusion index will be evaluated by recording the correlation between radial artery and invasive measurements and the perfusion indexes of both hands simultaneously with Masimo.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing liver transplantation Patients who will undergo intraarterial cannulation

Exclusion Criteria:

Peripheral vascular diseases Prior upper extremity surgery Radial artery injury

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the perfusion index of the hand in which artery cannulation was performed with Masimo.There is no result range | Intraoperative (patients during surgery)
  Arterial cannulation is mandatory for hemodynamic data monitoring in liver transplantation and is performed routinely. To evaluate the perfusion of the hand of the patients after cannulation

CONTACTS AND LOCATIONS:
Overall Officials: duygu demiröz, Principal Investigator — INONU UNİVERSİTY

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brzezinski M, Luisetti T, London MJ. Radial artery cannulation: a comprehensive review of recent anatomic and physiologic investigations. Anesth Analg. 2009 Dec;109(6):1763-81. doi: 10.1213/ANE.0b013e3181bbd416. PMID 19923502
- [Background] Numaguchi A, Adachi YU, Aoki Y, Ishii Y, Suzuki K, Obata Y, Sato S, Nishiwaki K, Matsuda N. Radial artery cannulation decreases the distal arterial blood flow measured by power Doppler ultrasound. J Clin Monit Comput. 2015 Oct;29(5):653-7. doi: 10.1007/s10877-014-9648-5. Epub 2014 Dec 16. PMID 25516161